CLINICAL TRIAL: NCT04899544
Title: Randomized Controlled Trial of Center-Based vs. In-Home Pivotal Response Treatment (PRT) in Autism
Brief Title: Trial of Center-Based vs. In-Home Pivotal Response Treatment (PRT) in Autism
Acronym: PRT-HvC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Anonymous Donor (Unknown)
Responsible Party: Principal Investigator, Antonio Hardan, Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-61427
Record Dates: First submitted 2021-05-19; First posted 2021-05-24 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Autism; Autism Spectrum Disorder; ASD
Keywords: pivotal response treatment; PRT; center based; social and communication
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder; Communication | interventions — Hypoxanthine Phosphoribosyltransferase; Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome raters and video coding rating are blinded to group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Center-Based Pivotal Response Treatment (PRT) Intervention (PRT-C) (Experimental): A 16-week center-based PRT intervention (PRT-C) consisting of 12 hours per week including 1 hour of parent training. This intervention targets social communication deficits.
  Interventions: Behavioral: Center-Based Pivotal Response Treatment (PRT) Intervention (PRT-C)
- Home-Based Pivotal Response Treatment (PRT) Intervention (PRT-H) (Experimental): A 16-week home-based PRT intervention (PRT-H) consisting of 12 hours per week including 1 hour of parent training. This intervention targets social communication deficits.
  Interventions: Behavioral: Home-Based Pivotal Response Treatment (PRT Intervention (PRT-H)
- Treatment As Usual (TAU) (No Intervention): This is a control group that consists of children who are receiving treatment as usual (TAU) for a 16-week period. These families will be invited to participate in PRT after completing the 16-week TAU phase.

INTERVENTIONS:
Behavioral: Center-Based Pivotal Response Treatment (PRT) Intervention (PRT-C) — Pivotal Response Treatment in autism center.
  Arms: Center-Based Pivotal Response Treatment (PRT) Intervention (PRT-C)
Behavioral: Home-Based Pivotal Response Treatment (PRT Intervention (PRT-H) — Pivotal Response Treatment in home environment.
  Arms: Home-Based Pivotal Response Treatment (PRT) Intervention (PRT-H)

SUMMARY:
The aim of this clinical trial is to compare the efficacy of a 16-week center-based Pivotal Response Treatment (PRT-C) versus home-based Pivotal Response Treatment (PRT-H) in targeting social communication deficits in young children with autism spectrum disorder (ASD) with significant language delay. The two groups will also be compared to a control group that consists of children who are receiving treatment as usual (TAU).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Autism Spectrum Disorder (ASD) based on Autism Diagnostic Interview Revised (ADI-R), Autism Diagnostic Observation Schedule, Second Edition (ADOS-2) or Childhood Autism Rating Scale, Second Edition (CARS-2), Diagnostic and Statistical Manual 5th Edition (DSM-5), and expert clinical opinion;
* Boys and girls between 2.0 and 5.11 years;
* Ability to participate in the testing procedures to the extent that valid standard scores can be obtained;
* Language delay as measured by the Preschool Language Scale, 5th Edition (PLS-5): Standard score at least 1 standard deviation below average for expressive language ability for 2 and 3 year olds; 2 standard deviations for 4 year olds, and 3 standard deviations for 5 year olds;
* Stable treatment (e.g., Applied Behavior Analysis - ABA), speech therapy, school placement, psychotropic medication(s) or biomedical intervention(s) for at least 1 month prior to baseline measurements;
* No anticipated changes on treatment during study participation for Center-Based Pivotal Response Treatment (PRT-C) and In-Home Pivotal Response Treatment (PRT-H);
* No more than 60 minutes of individual 1:1 speech therapy per week;
* Availability of at least one parent or primary caregiver who can consistently participate in parent training and research measures.

Exclusion Criteria:

* Current or lifetime diagnosis of severe psychiatric disorder (e.g., bipolar disorder, etc.);
* Receiving ABA of 15 hours or more;
* Presence of active medical problem (e.g., unstable seizure disorder or heart disease);
* Previous adequate Pivotal Response Treatment (PRT) trial;
* Participants living more than 30 miles from Stanford University;
* Child's primary language other than English.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2022-10-18 (Actual); Primary Completion 2028-09-15 (Estimated); Study Completion 2028-09-15 (Estimated)

PRIMARY OUTCOMES:
Change in Number of Child Utterances during the Parent-Child portion of the Structured Lab Observation (SLO). | Baseline,16 Weeks.

SECONDARY OUTCOMES:
Change on MacArthur-Bates Communication Development Inventory (CDI) Scores | Baseline,16 Weeks.
Change From Baseline in Parent Rated Vineland Adaptive Behavior Scale- 3 (VABS-3) Scores | Baseline,16 Weeks.
Change From Baseline in Parent Rated Social Responsiveness Scale, 2nd Edition (SRS-2) Scores | Baseline,16 Weeks.
  Social Responsiveness Scale, 2nd Edition (SRS-2) scores measure social abilities with lower scores meaning better social abilities.
Change From Baseline in Parent Rated Stanford Social Dimension Scale (SSDS) Scores | Baseline,16 Weeks.
  Higher Scores on the Stanford Social Dimension Scale mean better social functioning and lower scores mean worse social functioning (Range: 58-290).
Change on the Brief Observation of Social Communication Change (BOSCC) direct child observation assessment. | Baseline,16 Weeks.
Change on the Clinical Global Impressions (CGI) Scale. | Baseline,16 Weeks.

OTHER OUTCOMES:
Change From Baseline in the Parent Rated Emotion Dysregulation Inventory-Young Child (EDI-YC) Scores | Baseline,16 Weeks.
Change From Baseline in the Parent Rated General Self Efficacy Scale (GSES) Scores | Baseline,16 Weeks.
Change From Baseline in the Parent Rated Sensory Experiences Questionnaire (SEQ) Scores | Baseline,16 Weeks.
Change From Baseline in the Parent Rated Child and Family Quality of Life - 2 (CFQL-2) Scores | Baseline,16 Weeks.
Change From Baseline in the Parent Rated Behavior Rating Inventory of Executive Function-Preschool (BRIEF-P) Scores | Baseline,16 Weeks.
Change From Baseline in the Parent Rated Family Empowerment Scale (FES) Scores | Baseline,16 Weeks.
Change From Baseline in the Parent Rated Parent Motivation Inventory (PMI) Scores | Baseline,16 Weeks.
Change From Baseline in the Parent Rated Parent Stress Index, Short Form (PSI/SF) Scores | Baseline,16 Weeks.
Change From Baseline in the Parent Rated Dimensional Assessment of Repetitive Behaviors (DARB) Scores | Baseline,16 Weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Y. Hardan, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No